CLINICAL TRIAL: NCT03043820
Title: Raloxifene Augmentation in Patients With a Schizophrenia Spectrum Disorder to Reduce Symptoms and Improve Cognition
Brief Title: Raloxifene Augmentation in Patients With a Schizophrenia Spectrum Disorder
Acronym: RAPSODI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iris Sommer (Other)
Collaborators: Julius Center (Other); Rudolf Magnus Institute - University of Utrecht (Other); GGZ Eindhoven (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); GGZ Centraal (Other); Altrecht GGZ (Unknown); Reinier van Arkel Group (Unknown); Ziekenhuis Netwerk Antwerpen (ZNA) (Other)
Responsible Party: Sponsor-Investigator, Iris Sommer, Prof. dr. Iris Sommer, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL.55343.041.16; 2015-004483-11 (EudraCT Number); 80-83600-98-40120 (Other Grant/Funding Number: ZonMw)
Record Dates: First submitted 2016-10-25; First posted 2017-02-06 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder; Psychosis NOS
Keywords: raloxifene; selective estrogen receptor modulator (SERM); schizophrenia; psychosis; cognition; negative symptoms
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raloxifene (Active Comparator): Raloxifene 120 mg (2 tablets of 60mg) daily for 12 weeks.
  Interventions: Drug: Raloxifene
- Placebo (Placebo Comparator): Placebo 2 tablets daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Raloxifene — Oral selective estrogen receptor modulator (SERM).
  Other Names: Evista
  Arms: Raloxifene
Drug: Placebo — Tablets identical in form and color to intervention.
  Arms: Placebo

SUMMARY:
There is increasing clinical and molecular evidence for the role of hormones and specifically estrogen and its receptor in schizophrenia. A selective estrogen receptor modulator, raloxifene, stimulates estrogen-like activity in brain and can improve cognition in older adults. The present study will test the extent to which adjunctive raloxifene treatment improved cognition and reduced symptoms in young to middle-age men and women with schizophrenia.

110 patients with a schizophrenia spectrum disorder will be recruited in a multicenter twelve-week, randomized, double-blind, placebo-controlled, parallel trial of adjunctive 120mg raloxifene treatment in addition to their usual antipsychotic medications.

The investigators hypothesize that daily treatment with raloxifene 120 milligrams (mg) in addition to antipsychotic treatment improves cognition, reduces psychotic symptoms, increases social and personal functioning and reduces health care costs, as compared to placebo.

DETAILED DESCRIPTION:
Rationale:

Patients with a schizophrenia spectrum disorder experience substantial impairments in multiple domains of everyday life, including the ability to maintain social relationships, sustain employment, and live independently. These problems often persist, even after successful treatment of psychosis. Currently, no consistent evidence exists for the efficacy of interventions to reduce cognitive and negative symptoms, while in fact these are the factors that determine functioning to a great extent.

Premenopausal women with schizophrenia have less psychotic and negative symptoms, and better cognitive and social functioning, in comparison to men and older women. This has been related to protective effects of estrogens in the brain. Administering estrogens has positive effects on psychotic symptoms, but exerts long-term side effects, especially in men.

Raloxifene is a selective estrogen receptor modulator, with a beneficial side effect profile in women and in men. It has been shown to be effective in reducing symptoms in postmenopausal women with schizophrenia. Recently, positive results were found in premenopausal women and in men. It is important to replicate these results in an independent sample and to investigate the effects of raloxifene on functioning.

Hypotheses: Daily treatment with raloxifene 120 milligrams (mg) in addition to antipsychotic treatment improves cognition, reduces psychotic symptoms, increases social and personal functioning and reduces health care costs, as compared to placebo.

Objective:

The primary objective of this trial is to investigate the hypothesized beneficial effect of raloxifene as compared to placebo when given for twelve weeks in addition to antipsychotic medication to patients with a psychotic disorder. The investigators expect lower symptom severity as measured with the Positive And Negative Symptom Scale (PANSS) and improvements of cognitive functioning as measured with the Brief Assessment of Cognition in Schizophrenia (BACS).

Secondary objectives include reducement of negative symptoms as measured with the Brief Negative Symptom Scale (BNSS), improvement of Personal and Social Performance (using the PSP-scale), reduction of thought disorder symptoms measures with the Thought And Language Disorder-scale (TALD), reduction use of health care recourses using the institute for Medical Technology Assessment's Medical Consumption Questionnaire (iMTA-MCQ), productivity using the institute for Medical Technology Assessment's Productivity Cost Questionnaire (iMTA-PCQ), improvement of quality of life using the EuroQol-5 dimensions scale (EQ-5D), improvement in both speed and error rates in the Stroop test, reduction of comorbid depression using Beck's Depression Inventory (BDI), improvement of language production and various hormonal and inflammatory parameters.

Study design: Randomized placebo-controlled multicenter double-blind trial

Study population:

110 men and women diagnosed with schizophrenia, schizoaffective or schizophreniform disorder, or psychotic disorder not otherwise specified (DSM-IV 295.*)

Intervention:

Patients will be randomized 1:1 to either 120mg raloxifene or placebo daily for a period of 12 weeks. Identical tablets will be administered.

Main study parameters/endpoints:

Primary outcomes are changes in symptom severity as measured with PANSS and changes in cognition as measured with BACS. Secondary outcome are changes in negative symptoms (measured with BNSS), changes in personal and social performance (measured with PSP), change in severity of thought disorder (measured with TALD), quality of life (measured with EQ-5D), use of healthcare and non-healthcare resources, comorbid depression (measured with BDI), cognitive control (measured with a Stroop Test), language production (measured by analyzing speech samples) and hormonal and inflammatory biomarkers.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Use of raloxifene is associated with a small risk of side effects. The number of patient visits will be limited and mainly requires time invested for physical examinations, questionnaires and cognitive testing sessions (around 9 hours in total over the course of 9 months). Blood will be drawn at three occasions with negligible and known risks (e.g. irritation). The burden and risks are acceptable while the benefits are expected to be considerable.

ELIGIBILITY:
Inclusion Criteria:

* A DSM-IV-R diagnosis of: 295.x (schizophrenia, schizophreniform disorder, schizoaffective disorder, or psychotic disorder NOS)
* Capable of understanding the purpose and details of the study in order to provide written informed consent;
* On a stable dose of antipsychotic medication for at least two weeks;

For female patients:

* Female patients who are sexually active must be willing and capable to use a non-estrogenic contraceptive (intrauterine device, cervical cap, condom or diaphragm) in case of sexual intercourse for the complete duration of the study;
* Female patients with post coital uterine bleeding must have documented normal PAP smear and pelvic examination in the preceding two years.

Exclusion Criteria:

* Pre-existing cardiovascular disease;
* History of thrombo-embolic events;
* History of breast cancer;
* Familial tendency to form blood clots (such as familial factor V Leiden);
* Use of vitamin K antagonists;
* Use of cholestyramine or other anion exchange resins;
* Hypertriglyceridemia (triglycerides > 3 times the upper limit of normal (ULN));
* Liver function or enzyme disorders (serum bilirubin, alkaline phosphatase (AF), gamma-glutamyl transpeptidase (γ - GT), aspartate aminotransferase (ASAT) or alanine aminotransferase (ALAT) > 3 times the ULN as measured at baseline);
* Severe kidney failure (eGFR <30 ml/min as measured at baseline);
* Use of any form of estrogen, progestin or androgen as hormonal therapy, or antiandrogen including tibolone or use of phytoestrogen supplements as powder or tablet in the past three months.

For female patients:

* Abnormality observed during physical breast examination;
* Pregnancy or breast feeding;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Change in symptom severity as measured with the Positive and Negative Symptom Scale (PANSS) | Baseline, at 6 weeks of treatment, at 12 weeks of treatment (end of treatment) and 6 months after end of treatment (follow-up)
  Effect of the study therapies on symptom severity.
Change in cognitive functioning as measured with the Brief Assessment of Cognition in Schizophrenia | Baseline, at 12 weeks (end of treatment) and 6 months after end of treatment (follow-up)
  Effect of the study therapies on cognitive functioning

SECONDARY OUTCOMES:
Personal and social performance measured with the Personal and Social Performance scale (PSP) | Baseline, at 6 weeks, at 12 weeks (end of treatment) and 6 months after end of treatment (follow-up)
  Effect of the study therapy on personal and social performance.
Thought disorder severity as measured with the Thought And Language Disorder scale (TALD) | Baseline, at 6 weeks, at 12 weeks (end of treatment) and 6 months after end of treatment (follow-up)
  Effect of the study therapy on severity of thought disorder.
Participant's Quality of Life as measured with the EQ-5D-5L | Baseline, at 12 weeks (end of treatment) and 6 months after end of treatment (follow-up)
  Effect of the study therapy on quality of life.
Comorbid depression as measured with Beck's Depression Inventory (BDI). | Baseline, at 6 weeks, at 12 weeks (end of treatment) and 6 months after end of treatment (follow-up)
  Effect of the study therapy on comorbid depression
Use of health-recourses as measured with the iMTA-MCQ | Baseline, at 12 weeks (end of treatment) and 6 months follow-up
  Effect of the study therapy on use of recourses.
Use of non-health recourses as measured with the iMTA-PCQ | Baseline, at 12 weeks (end of treatment) and 6 months after end of treatment (follow-up)
  Effect of the study therapy on use of recourses.
Language production assessment by analyzing speech samples | Baseline and at 12 weeks of treatment (end of treatment)
  Effect of the study therapy on free speech.
Symptom severity as measured with the Brief Negative Symptom Scale (BNSS) | Baseline, at 6 weeks, at 12 weeks (end of treatment) and 6 months after end of treatment (follow-up)
  Effect of the study therapies on symptom severity.

OTHER OUTCOMES:
Hormonal biomarkers for predicting treatment response to raloxifene | Baseline and at 12 weeks of treatment
  Hormonal biomarkers (in women: prolactin, follicle stimulating hormone and 17-beta estradiol; in men: prolactin, 17-beta estradiol, testosterone and sex hormone binding globulin and c-reactive protein will be assessed in blood samples to examine whether these parameters predict treatment response to raloxifene augmentation.
Deoxyribonucleic acid analysis for predicting treatment response to raloxifene | Baseline and at 12 weeks of treatment
  Single nucleotide polymorphism (SNP) analysis of estrogen receptor gene 1 (ESR1) SNP rs2234693, rs9340799, rs2144025 and UGT1A8 gene rs1042597.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Sommer, Prof. dr., Principal Investigator — UMC Groningen; Bob Oranje, Ass. Prof., Principal Investigator — UMC Utrecht; Janna de Boer, MD, Study Chair — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Heringa SM, Begemann MJ, Goverde AJ, Sommer IE. Sex hormones and oxytocin augmentation strategies in schizophrenia: A quantitative review. Schizophr Res. 2015 Nov;168(3):603-13. doi: 10.1016/j.schres.2015.04.002. Epub 2015 Apr 23. PMID 25914107